CLINICAL TRIAL: NCT04270942
Title: An Open-Label Study to Evaluate the Safety of Teplizumab (PRV-031) in At-Risk Relatives Who Develop Type 1 Diabetes
Brief Title: At-Risk for Type 1 Diabetes Extension Study (TN-10 Extension)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Provention Bio, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRV-031-002; SFY18115 (Other: Sanofi Identifier)
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Recent-onset type 1 diabetes; Teplizumab; T1D; Stage 3; Type 1 diabetes; New onset type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — teplizumab

STUDY DESIGN:
Intervention Model Description: Single-arm, multicenter, open-label clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Teplizumab treated (Experimental): Administration of teplizumab by intravenous infusion for 12 consecutive days
  Interventions: Drug: teplizumab 1 mg/mL

INTERVENTIONS:
Drug: teplizumab 1 mg/mL — Solution for infusion administered as IV infusion (anti-CD3 humanized monoclonal antibody).
  Cumulative dose: 9 mg/m2. Day 1: 106 μg/m2, Day 2: 425 μg/m2, Days 3-12: 850 μg/m2 daily
  Other Names: PRV-031, Tzield

SUMMARY:
This study was an extension of the NIH-sponsored At-Risk (TN-10) type 1 diabetes study (NCT 01030861). Teplizumab-treated and placebo-treated participants in the NIH trial who developed clinical type 1 diabetes after the conclusion of that trial, were eligible to enroll and receive teplizumab treatment within one year of diagnosis of clinical type 1 diabetes.

DETAILED DESCRIPTION:
The study was a single-arm, multicenter, open-label clinical trial. All participants received a 12-day course of teplizumab given through daily IV infusion and were followed for 78 weeks.

The purpose of this study was to evaluate the safety and tolerability of teplizumab treatment, administered intravenously (IV) to participants in the NIH-sponsored trial who have developed type 1 diabetes and were able to start teplizumab treatment within 1 year of diagnosis of type 1 diabetes. Whether teplizumab treatment reduced the loss of insulin-producing pancreatic beta cells were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Previous participant in the TN-10 study
2. Participant had received a diagnosis of type 1 diabetes after the conclusion of the TN-10 study, according to the criteria from the American Diabetes Association (ADA).
3. Participant was able to initiate teplizumab treatment required in this study within 1 year of type 1 diabetes diagnosis.
4. Participant was willing to forego other forms of experimental treatment during the entire study.
5. Participant and/or guardian had given informed consent and assent as applicable.

Exclusion Criteria:

1. Had an active infection and/or fever.
2. Had a history of or serologic evidence at screening of current or past infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
3. An individual who had a medical, psychological or social condition that, in the opinion of the Principal Investigator, would interfere with safe and proper completion of the trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (8):
- United States (8):
  - Barbara Davis Center for Diabetes Site Number : 04, Aurora, Colorado
  - Clinical Site, Aurora, Colorado
  - Yale University School of Medicine Site Number : 01, New Haven, Connecticut
  - Clinical Site, New Haven, Connecticut
  - Clinical Site, Gainesville, Florida
  - University of Florida Site Number : 02, Gainesville, Florida
  - Clinical Site, Nashville, Tennessee
  - Vanderbilt Univerity Medical Center Site Number : 03, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in the United States from 26-Feb-2020 to 22-Jan-2024.
Pre-assignment Details: A total of 6 participants from the TN-10 study (NCT01030861) who developed clinical (stage 3) type 1 diabetes (T1D) after the completion of that study were enrolled in this study. All participants received teplizumab in this study within 1 year of diagnosis of clinical T1D.
Groups:
- Teplizumab: Participants received teplizumab 9 milligrams per meter square (mg/m^2) via intravenous (IV) infusion as a 12-day course (once daily) split as: Day 1: 106 micrograms (mcg)/m^2, Day 2: 425 mcg/m^2 and Days 3 to 12: 850 mcg/m^2.
Period: Overall Study
Arm/Group | Teplizumab
Started | 6
Completed | 5
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of teplizumab.
Groups:
- Teplizumab: Participants received teplizumab 9 mg/m^2 via IV infusion as a 12-day course (once daily) split as: Day 1: 106 mcg/m^2, Day 2: 425 mcg/m^2 and Days 3 to 12: 850 mcg/m^2.
Arm/Group | Teplizumab
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.3 (11.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Treatment-emergent Adverse Events of Special Interest (TEAESIs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant,temporally associated with use of study dose,whether or not considered related to study dose.AESI was any AE that met any of following:All >=Grade 3 infections (including all opportunistic infections);acute mononucleosis-like illness;lymphomas or other malignancies;severe hypoglycemic episode;>=Grade 3 liver function abnormalities, thrombocytopenia, neutropenia or rash;>= Grade 4 allergic/hypersensitivity reaction (anaphylaxis) or cytokine-release syndrome; lymphocyte count <500/cubic millimeter for 7 days or longer. An SAE was as any untoward medical occurrence that,at any dose:resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization,resulted in persistent disability/incapacity, was a congenital anomaly/birth defect or any other medically important event.A TEAE was any AE which started during or after the first dose of teplizumab.
Time Frame: From the first dose of study drug administration (Day 1) up to approximately 78 weeks
Population: The safety analysis set included all participants who received at least 1 dose of teplizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Teplizumab
Number analyzed (Participants) | 6
Participants
  Any TEAE | 6
  Any TEAESI | 0
  Any TESAE | 1

2. Secondary Outcome: Serum Concentration Immediately Prior to Administration of the Next Dose (Ctrough) of Teplizumab at Day 364
Description: Blood samples were collected for evaluation of pharmacokinetic (PK) data.
Time Frame: Pre-dose on Day 364
Population: The PK analysis set included all participants in the safety analysis set who had at least 1 eligible PK sample for analysis. Only those participants with data collected on Day 364 are reported.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Teplizumab
Number analyzed (Participants) | 5
nanogram/milliliter (ng/mL) | NA (NA) — NA indicates that Mean and Standard deviation could not be determined as the values were below the lower limit of quantification (LLOQ). LLOQ value was 2.50 ng/mL.

3. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) Against Teplizumab
Description: Blood samples were collected for the evaluation of ADA against teplizumab.
Time Frame: Up to Day 364
Population: The immunogenicity analysis set included all participants in the safety analysis set who had at least 1 eligible immunogenicity sample for analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Teplizumab: Participants received teplizumab 9 mg/m^2 via IV infusion as a 12-day course split as: Day 1: 106 mcg/m^2, Day 2: 425 mcg/m^2 and Days 3 to 12: 850 mcg/m^2.
Arm/Group | Teplizumab
Number analyzed (Participants) | 6
Participants | 6

4. Secondary Outcome: Area Under the Time-Versus-Concentration Curve (AUC) of C-peptide After a 4-hour (4h) Mixed Meal Tolerance Test (MMTT) at Week 78
Description: The AUC of C-peptide was measured after a 4-hour MMTT as a measure of assessing endogenous insulin production and beta cell function. The AUC was computed using the trapezoidal rule and standardized by the duration of the MMTT test for the analysis.
Time Frame: Week 78
Population: The safety analysis set included all participants who received at least 1 dose of teplizumab. Only those participants with data collected at Week 78 are reported.
Measure: Mean (Standard Deviation); unit: ln(AUC+1) (picomole/mL)
Arm/Group | Teplizumab
Number analyzed (Participants) | 4
ln(AUC+1) (picomole/mL) | 0.549 (0.4276)

5. Secondary Outcome: Glycated Hemoglobin (HbA1c) Levels at Week 78
Description: Blood samples were collected for evaluation of HbA1c.
Time Frame: Week 78
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Teplizumab
Number analyzed (Participants) | 4
percentage of HbA1c | 8.50 (3.785)

6. Secondary Outcome: Average Daily Use of Exogenous Insulin at Week 78
Description: The average daily insulin use was calculated based on participants who had at least 3 days of insulin use recorded in the diary for the Week 78 visit.
Time Frame: Week 78
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: unit/kilogram/day
Arm/Group | Teplizumab
Number analyzed (Participants) | 4
unit/kilogram/day | 0.54 (0.357)

7. Secondary Outcome: Number of Participants With Severe Hypoglycemic Episodes
Description: The severity of a hypoglycemia event was identified by the Investigator and classified according to National Cancer Institute-Common Terminology Criteria for Adverse Events version 5.0 as follows:
  * Grade 3 hypoglycemia: 30-39 milligram/deciliter (mg/dL) (1.7-2.1 millimole [mmol]/L). This is considered severe or medically significant but not immediately life-threatening. Hospitalization or prolongation of hospitalization is likely indicated. It is considered disabling and limits self-care.
  * Grade 4 hypoglycemia: <=29 mg/dL (1.6 mmol/L). This is considered life threatening (seizures) with urgent intervention indicated.
  * Grade 5 hypoglycemia: Hypoglycemia resulting in death. Hypoglycemia >=Grade 3 was considered as severe hypoglycemia.
Time Frame: From the first dose of study drug administration (Day 1) up to approximately 78 weeks
Population: The safety analysis set included all participants who received at least 1 dose of teplizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Teplizumab
Number analyzed (Participants) | 6
Participants | 0

8. Secondary Outcome: Number of Participants With Change in Cluster of Differentiation (CD)8+ TIGIT+ KLRG1+ T Cells
Description: CD8+ TIGIT+ KLRG1+ T cells were measured using flow cytometry.
Time Frame: From the first dose of study drug administration (Day 1) up to approximately 78 weeks
Population: The safety analysis set included all participants who received at least 1 dose of teplizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Teplizumab
Number analyzed (Participants) | 6
Participants | 4

ADVERSE EVENTS:
Time Frame: From the first dose of study drug administration (Day 1) up to approximately 78 weeks
Description: The safety analysis set included all participants who received at least 1 dose of teplizumab.
Arm/Group | Teplizumab
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teplizumab (N=6)
Completed Suicide (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teplizumab (N=6)
Leukopenia (Blood and lymphatic system disorders) | 2 (6)
Lymphopenia (Blood and lymphatic system disorders) | 3 (12)
Neutropenia (Blood and lymphatic system disorders) | 1 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (5)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Feeling Hot (General disorders) | 1 (2)
Infusion Site Pruritus (General disorders) | 1 (1)
Pain (General disorders) | 1 (2)
Pyrexia (General disorders) | 2 (2)
Cytokine Release Syndrome (Immune system disorders) | 1 (2)
Covid-19 (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (1)
Blood Lactate Dehydrogenase Increased (Investigations) | 1 (1)
Eosinophil Count Increased (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (10)
Neuralgia (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Rash Macular (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT04270942/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT04270942/SAP_001.pdf